CLINICAL TRIAL: NCT03894735
Title: The Effect of Serum Vitamin D and Calcium Levels in Ectopic Pregnancies
Brief Title: Vitamin D in Ectopic Pregnancies
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Principal investigator, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.08.11
Record Dates: First submitted 2019-03-27; First posted 2019-03-28 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Ectopic Pregnancy; Vitamin D Deficiency
Keywords: Calcium; Magnesium; Inflammation
MeSH Terms: conditions — Pregnancy, Ectopic; Vitamin D Deficiency; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to recent evidences, vitamin D was found to have important roles in female reproductive system, both in physiological and also pathological mechanisms. Since vitamin D is tightly related with calcium metabolism, both molecules were reported to be associated with some pregnancy complications including preeclampsia, gestational diabetes, low birth weight, preterm delivery, and cesarean section rates. The aim of the present study was to evaluate the vitamin D levels in ectopic pregnancies, which may have clinical importance in the etiology of this disorder.

ELIGIBILITY:
Inclusion Criteria:

* ectopic pregnancies and
* women with normal 1st trimester pregnancies

Exclusion Criteria:

* Patients without any known operations or
* disease history

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: ectopic pregnancies and women with normal 1st trimester pregnancies
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
vitamin D level | at the time of diagnosis of ectopic pregnancy
  vitamin d level value will be evaluated in ectopic pregnancies. 25-OH vitamin D (ng / ml) will be looked at in terms of vitamin levels.
vitamin D level | first trimester
  vitamin d level value will be evaluated in first trimester. 25-OH vitamin D (ng / ml) will be looked at in terms of vitamin levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)